CLINICAL TRIAL: NCT01296282
Title: Comparison Between Internal and External Chest Impedance Measurement
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Dr. Mark Kazatsker, Hillel Yaffe Medical Center
Other Study IDs: 0094-10-HYMC
Record Dates: First submitted 2011-02-13; First posted 2011-02-15 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Heart failure patients
  Interventions: Device: Medronics CRT Optivol Impedance Measurement; Device: External Thoracic Impedance Measurement

INTERVENTIONS:
Device: Medronics CRT Optivol Impedance Measurement — Pacemaker
Device: External Thoracic Impedance Measurement

SUMMARY:
To compare two methods of chest impedance: the Medtronics Optivol Measurement via CRT pacemakers for patients with heart failure and external non-invasive measurement

ELIGIBILITY:
Inclusion Criteria:

* CRT-implanted patients with heart failure

Exclusion Criteria:

* All others

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with heart failure with CRT pacemaker
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-03; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
External measurement of chest impedance can be effective in monitoring heart failure patients | Three years

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel